CLINICAL TRIAL: NCT03444753
Title: A Phase I Study of BMS-986299 as Monotherapy and in Combination With Nivolumab and Ipilimumab in Participants With Advanced Solid Cancers
Brief Title: An Investigational Immunotherapy Study of BMS-986299 Alone and in Combination With Nivolumab and Ipilimumab in Participants With Solid Cancers That Have Spread or Cannot be Removed
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA039-001
Record Dates: First submitted 2018-02-20; First posted 2018-02-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): BMS-986299
  Interventions: Drug: BMS-986299
- Arm B (Experimental): BMS-986299 in combination with nivolumab and ipilimumab
  Interventions: Drug: BMS-986299; Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Drug: BMS-986299 — Specified dose on specified day
Biological: Nivolumab — Specified dose on specified day
  Other Names: Opdivo; BMS-936558
  Arms: Arm B
Biological: Ipilimumab — Specified dose on specified day
  Other Names: Yervoy; BMS-734016
  Arms: Arm B

SUMMARY:
The purpose of this study is to determine whether BMS-986299 both by itself and in combination with Nivolumab and Ipilimumab is safe and tolerable in the treatment of advanced solid tumors. In addition, the ability of study drugs to stimulate an immune response against cancer will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced/metastatic solid tumor and refractory to or intolerant of existing therapy(ies) known to provide clinical benefit for the condition of the participant
* IO therapy resistant or insensitive tumors
* Have at least 2 tumor lesions accessible for biopsy
* Eastern Cooperative Oncology Group Performance Status of 0 or 1

Exclusion Criteria:

* Primary CNS malignancy
* Participants with other active malignancy requiring concurrent intervention
* Uncontrolled or significant cardiovascular disease

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | Up to 28 days
Incidence of adverse events (AEs) | Approximately 2 years
Incidence of clinical laboratory abnormalities | Approximately 2 years
Incidence of serious adverse events (SAEs) | Approximately 2 years
Incidence of AEs leading to discontinuation and deaths | Approximately 2 years

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Approximately 2 years
Time of maximum observed plasma concentration (Tmax) | Approximately 2 years
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] | Approximately 2 years
Area under the plasma concentration-time curve from time zero to 24 hours postdose [AUC(0-24)] | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- United States (9):
  - Local Institution - 0003, La Jolla, California
  - Local Institution, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - Local Institution, New Haven, Connecticut
  - Local Institution, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Local Institution, Portland, Oregon
  - Local Institution, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Nelson BE, O'Brien S, Sheth RA, Hong DS, Naing A, Zhang X, Xu A, Hamuro L, Suryawanshi R, McKinley D, Novosiadly RD, Piha-Paul SA. Phase I study of BMS-986299, an NLRP3 agonist, as monotherapy and in combination with nivolumab and ipilimumab in patients with advanced solid tumors. J Immunother Cancer. 2025 Jan 16;13(1):e010013. doi: 10.1136/jitc-2024-010013. PMID 39824531
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/safety/medwatch/safetyinformation/default.htm